CLINICAL TRIAL: NCT05293015
Title: NP-Supported Multidisciplinary Diabetes Management During Perioperative Period in Patient With Diabetes Mellitus
Brief Title: NP-Supported Multidisciplinary Diabetes Management During Perioperative Period
Acronym: NPMDM-PP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M2021609
Record Dates: First submitted 2021-12-29; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-12

CONDITIONS: Diabetes
Keywords: nurse practitioners, Multidisciplinary Diabetes Management, perioperative period
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NP-Supported Multidisciplinary Diabetes Management (Experimental): NP establishes files to evaluate and manage patients before hospital and visits patients after hospitalization. Then set blood glucose control goals with endocrinology and orthopedic doctors together, initiates consultation with endocrinologists for patients with postoperative hyperglycemia, and is responsible for post-hospital follow-up.
  Interventions: Other: NP-Supported Multidisciplinary Diabetes Management
- Regular diabetes management (No Intervention): The patient would go to the endocrinology outpatient clinic before hospitalization to regulate blood glucose, and be managed by by orthopedic medical staff through hospitalization. If necessary, the endocrinologist is consulted. And after the hospital, patients would be followed up by orthopedic medical staff.

INTERVENTIONS:
Other: NP-Supported Multidisciplinary Diabetes Management — NP establishes files to evaluate and manage patients before hospital and visits patients after hospitalization. Then set blood glucose control goals with endocrinology and orthopedic doctors together, initiates consultation with endocrinologists for patients with postoperative hyperglycemia, and is responsible for post-hospital follow-up.
  Arms: NP-Supported Multidisciplinary Diabetes Management

SUMMARY:
The primary objective of this study is to determine the benefits of interventions from a Multidisciplinary Diabetes Care team involved of diabetes nurse practitioners(DNP) on glucose control, perioperative outcomes and psychosocial outcomes for patients with Diabetes Mellitus

DETAILED DESCRIPTION:
About 50% of diabetic patients will undergo at least one surgical operation, and nearly 20% of surgical patients have diabetes.Compared with non-diabetic patients, diabetic patients face greater risks during the perioperative period. Stress factors such as preoperative preparation, anesthesia, surgical trauma, pain, drugs and negative emotions can induce blood glucose fluctuations, which could lead to complications such as hyperglycemia, diabetic ketosis, and hypoglycemia.Therefore, perioperative management has become an important part of diabetes management.

A multidisciplinary collaborative team led by NP can reduce the mortality of patients after inpatient surgery, help patients change their lifestyle, maintain self-management behavior, improve patient experience, and reduce hospitalization costs. This study intends to explore the application effect of NP-led multidisciplinary collaborative team in the perioperative comprehensive management of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis meets World Health Organization (WHO) (1999) Diabetes Diagnostic Standards
* Orthopedic assessment requires elective surgery and no surgical contraindications
* HbA1c≥8.5% or intravenous fasting blood glucose (FBG)>10mmol/l
* Informed consent.

Exclusion Criteria:

* Cognitive and communication disorders;
* Pregnancy;
* Participate in other intervention studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: TIR（Time in Range） | From into the group to the first hospital day; First day in hospital to the day of discharge
  Time in range

SECONDARY OUTCOMES:
EFFICACY: Glycated Serum Protein | baseline and 1 month after discharged
  Glycated Serum Protein would be conducted to measure glucose control
EFFICACY: Incidence of perioperative hypoglycemia | From into the grop to 1 month after surgery. And confirmed based on the patient's main complaint and monitoring records.
  Incidence of perioperative hypoglycemia would be conducted to measure glucose control
EFFICACY: Time required for blood glucose standard before surgery | the first hospital day
  The time from the patient's enrollment to the blood glucose reaching the blood glucose control target
EFFICACY: Diabetes self-management behavior | Measurements were taken at baseline, day of hospitalization, and 1 month after discharge
  measured by Summary of Diabetes Self-Care Activities（SDSCA）. SDSCA scores from 0 to 77 and higher score means better self-management behaviors.
EFFICACY: Incidence of perioperative adverse events | 1 month after discharge
  Adverse events included wound infection, prolonged wound healing time, and death within 1 month after surgery.
EFFICACY: Blood pressure | baseline, day of hospitalization, during hospitalization and 1 month after discharge
  A calibrated electronic blood pressure meter of the same brand was used to measure systolic pressure and diastolic pressure in the same arm at the same time daily
EFFICACY: Body weight | baseline, day of hospitalization, during hospitalization and 1 month after discharge
  The same scale was used to measure after patients got up in the morning.
EFFICACY: Anxiety and depression | Measurements were taken at baseline, day of hospitalization, and 1 month after discharge
  measured by Hospital Anxiety and Depression Scale (HADS) scale. HADS contains two subscales: anxiety and depression, and each subscale have 7 items. Total scores were from 0 to 42(anxiety: 21 scores; depression: 21 scores), higher score means more severe anxiety and/or depression.
QUALITY OF LIFE:living quality | Measurements were taken at baseline, day of hospitalization, and 1 month after discharge
  measured by Short Form 36 Health Survey (SF-36) which contains 8 modules with different score formula. Higher total scores mean better living quality.

REFERENCES:
- [Background] Liao CC, Lin CS, Shih CC, Yeh CC, Chang YC, Lee YW, Chen TL. Increased risk of fracture and postfracture adverse events in patients with diabetes: two nationwide population-based retrospective cohort studies. Diabetes Care. 2014 Aug;37(8):2246-52. doi: 10.2337/dc13-2957. Epub 2014 May 7. PMID 24804698
- [Background] Meneghini LF. Perioperative management of diabetes: translating evidence into practice. Cleve Clin J Med. 2009 Nov;76 Suppl 4:S53-9. doi: 10.3949/ccjm.76.s4.09. PMID 19880837
- [Background] Clement S, Braithwaite SS, Magee MF, Ahmann A, Smith EP, Schafer RG, Hirsch IB; American Diabetes Association Diabetes in Hospitals Writing Committee. Management of diabetes and hyperglycemia in hospitals. Diabetes Care. 2004 Feb;27(2):553-91. doi: 10.2337/diacare.27.2.553. No abstract available. PMID 14747243
- [Background] Sebranek JJ, Lugli AK, Coursin DB. Glycaemic control in the perioperative period. Br J Anaesth. 2013 Dec;111 Suppl 1:i18-34. doi: 10.1093/bja/aet381. PMID 24335396
- [Background] Aminian A, Kashyap SR, Burguera B, Punchai S, Sharma G, Froylich D, Brethauer SA, Schauer PR. Incidence and Clinical Features of Diabetic Ketoacidosis After Bariatric and Metabolic Surgery. Diabetes Care. 2016 Apr;39(4):e50-3. doi: 10.2337/dc15-2647. Epub 2016 Jan 28. No abstract available. PMID 26822327
- [Background] Golden SH, Peart-Vigilance C, Kao WH, Brancati FL. Perioperative glycemic control and the risk of infectious complications in a cohort of adults with diabetes. Diabetes Care. 1999 Sep;22(9):1408-14. doi: 10.2337/diacare.22.9.1408. PMID 10480501